CLINICAL TRIAL: NCT01666964
Title: Prevalence of Hypopituitarism Following Combat-related Traumatic Brain Injury in a Military Population
Brief Title: Hormone Deficiency After Brain Injury During Combat
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 350758-12
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Traumatic Brain Injury; Hypopituitarism
Keywords: Traumatic brain injury; hypopituitarism
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypopituitarism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No specimens will be stored.
  Blood Testing:
  Testosterone 2ml Estradiol 2ml LH/FSH 3ml Prolactin 2ml IGF-1 1ml TSH 2ml Free T4 1ml Sodium 2ml Total blood for cosyntropin stim test 9ml Total blood for glucagon stim test 15ml Water deprivation testing 12ml-32ml
  Urine Testing:
  HCG 2ml Water deprivation testing 8ml-18ml
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 3 months post-injury: Male and female combat veterans age 18 years and older with the diagnosis of Traumatic Brain Injury caused by a blast that occurred 3 months prior to enrollment, 50% mild, 50% moderate and severe
  Interventions: Other: Blast Traumatic Brain Injury
- 6 months post-injury: Male and female combat veterans age 18 years and older with the diagnosis of Traumatic Brain Injury caused by a blast that occurred 6 months prior to enrollment, 50% mild, 50% moderate and severe
  Interventions: Other: Blast Traumatic Brain Injury

INTERVENTIONS:
Other: Blast Traumatic Brain Injury — Exposure during combat to blast-wave mediated Traumatic Brain Injury
  Other Names: bTBI

SUMMARY:
We would like to ascertain the prevalence of hypopituitarism after combat-related TBI. This will lead to enhanced awareness, recognition, and treatment of hypopituitarism, which can have life-saving ramifications and enhance quality of life and rehabilitation efforts in our combat veterans.

DETAILED DESCRIPTION:
The prevalence of hypopituitarism after combat-related traumatic brain injury (TBI) is currently unknown. Recent civilian data on TBI show the prevalence of any pituitary hormone deficiency is as high as 80% after 12 months. While the military prevalence of hypopituitarism can be extrapolated from civilian data, a major limitation is the notably different mechanism of injury (i.e., blast) for military personnel compared to civilians (i.e., assaults, traffic accidents and falls). Little is known about the effect of shockwaves from a blast injury on central nervous system tissue, and due to the unique nature of blast-related TBI, the prevalence of pituitary dysfunction in affected service members may significantly differ from nonmilitary subjects in prior studies.

ELIGIBILITY:
Inclusion Criteria:

* Combat veterans who are 3 or 6 months post combat-related TBI and age 18yrs or older
* Must demonstrate capacity for informed consent
* Must be DEERS eligible (Military healthcare beneficiary)

Exclusion Criteria:

* Pregnancy (to be assessed by urine HCG)
* Use of hormonal contraceptives
* Chronic oral or intravenous glucocorticoids
* Use of hormonal therapy to include estrogen and testosterone
* Prior diagnosis of hypopituitarism prior to combat related TBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female combat veterans age 18 years and older with the diagnosis of Traumatic Brain Injury that occurred 3 and 6 months prior to enrollment.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anterior pituitary dysfunction | at 3 (+/- 15 days) and 6 months (+/- 15 days)
  Pituitary screening blood tests: cortisol, follicle stimulating hormone, luteinizing hormone, total testosterone (males) or estradiol (females), thyrotropin, free thyroxine, prolactin, insulin-like growth factor-1. Growth-hormone deficiency will be confirmed with a glucagon stimulation test. Adrenal Insufficiency will be confirmed with an Cosyntropin stimulation test.

SECONDARY OUTCOMES:
Prevalence of posterior pituitary dysfunction | at 3 and 6 months
  Pituitary Dysfunction: Screening Sodium. Diabetes Insipidus will be confirmed with a water deprivation test.

OTHER OUTCOMES:
Background prevalence of hypopituitarism in a military population using the Department of Defense serum repository | At completion of Enrollment
  Screening labs for pituitary dysfunction repeated on frozen serum obtained prior to injury.
Relationship between hypopituitarism secondary to combat-related TBI and symptom scores using the Neurobehavioral Symptom Index. | 3 and 6 months post-injury
  The Neurobehavioral Symptom Index is a validated measure of cognitive and somatic symptoms after Traumatic Brain Injury.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Brackbill, M.D., Principal Investigator — WalterReed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States